CLINICAL TRIAL: NCT03924193
Title: Cognitive-Behavioral and Pharmacologic (LDX) Treatment of Binge-Eating Disorder and Obesity
Brief Title: Cognitive-Behavioral and Pharmacologic (LDX) Treatment of Binge-Eating Disorder and Obesity: Acute Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000022480_b; 1R01DK114075-01A1 (NIH)
Record Dates: First submitted 2019-04-17; First posted 2019-04-23 (Actual); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Binge-Eating Disorder; Obesity
MeSH Terms: conditions — Binge-Eating Disorder; Obesity | interventions — Lisdexamfetamine Dimesylate; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LDX (Active Comparator)
  Interventions: Drug: Lisdexamfetamine Dimesylate
- Cognitive-Behavioral Therapy (Active Comparator)
  Interventions: Behavioral: Cognitive-Behavioral Therapy
- LDX and Cognitive Behavioral Therapy (Active Comparator)
  Interventions: Other: Combination LDX and Cognitive-Behavioral Therapy

INTERVENTIONS:
Drug: Lisdexamfetamine Dimesylate — Participants randomly assigned to this arm will receive 12 weeks of LDX medication.
  Arms: LDX
Behavioral: Cognitive-Behavioral Therapy — Participants randomly assigned to this arm will receive 12 weeks of Cognitive-Behavioral Therapy
  Arms: Cognitive-Behavioral Therapy
Other: Combination LDX and Cognitive-Behavioral Therapy — Participants randomly assigned to this arm will receive 12 weeks of LDX and Cognitive-Behavioral Therapy
  Arms: LDX and Cognitive Behavioral Therapy

SUMMARY:
Brief Summary: This study will compare the effectiveness of cognitive behavioral therapy (CBT), lisdexamfetamine (LDX), and the combination of CBT and LDX for the treatment of binge-eating disorder in patients with obesity. This is an acute treatment comparing CBT or LDX alone or in combination.

DETAILED DESCRIPTION:
Obesity is a heterogeneous problem and research has highlighted the particular significance of a subgroup with binge-eating disorder (BED), the most prevalent formal eating disorder. This study examined the effectiveness of two leading but distinct treatments - lisdexamfetamine (LDX) and cognitive behavioral therapy (CBT) - alone and in combination, for BED in patients with obesity. LDX is the first and only FDA-approved medication for the treatment of BED and has demonstrated short-term effectiveness relative to placebo. CBT is the best-established psychological treatment, has demonstrated short-term effectiveness and "treatment specificity" (i.e., superiority to a variety of control and active treatments), has shown longer-term superiority to fluoxetine, and longer-term durability of outcomes. N=180 participants with BED and obesity will be randomly assigned to one of three interventions, CBT alone, LDX alone, or CBT combined with LDX. This RCT will provide new findings regarding the relative effectiveness of LDX, CBT, and combined CBT+LDX for patients with obesity and BED. No such study has been performed.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 64 years old
* Meets DSM-5 criteria for binge-eating disorder
* BMI 27-30 with a controlled obesity-related co-morbidity; or BMI ≥ 30 and <50
* Medically cleared as determined by EKG and medical record review
* Available for the duration of the treatment and follow-up (18 months)
* Read, comprehend, and write English at a sufficient level to complete study-related materials
* Able to travel to study location (New Haven, CT) for weekly visits

Exclusion Criteria:

* Previous history of problems with LDX or other stimulants
* Current psychostimulant use or use of any medication for ADHD
* Current use of study medications: LDX (Vyvanse), Bupropion (Wellbutrin, Zyban), Naltrexone, or Contrave
* History of congenital heart disease, known structural cardiac abnormalities, cardiomyopathy, serious heart arrhythmia, coronary artery disease, cerebrovascular pathology including stroke, exertional chest pain, uncontrolled high blood pressure, and other serious heart problems.
* History of severe renal, hepatic, neurological, or chronic pulmonary disease or other serious, unstable medical disorder.
* Current uncontrolled hypertension
* Current uncontrolled type I or II diabetes mellitus
* Current uncontrolled thyroid illness
* Gallbladder disease
* Co-occurring severe mental illness requiring hospitalization or intensive treatment
* Endorses current active suicidal or homicidal ideation with intent or plan
* History or current alcohol or substance use disorder (smoking is not exclusionary)
* Predisposition to seizures
* History of anorexia nervosa or bulimia nervosa, or currently regularly self-inducing vomiting
* Currently taking MAOI, SSRI or strong inhibitors of CYP2D6
* History of allergy or sensitivity to the study medication or stimulant medications
* Current use of medications contraindicated with the study medications
* Currently breast feeding or pregnant, or not willing to use reliable form of contraception
* Currently taking opioid pain medications or drugs
* Currently using effective treatment (evidence-based therapeutic or psychopharmacologic) for eating and/or weight loss
* Currently participating in another clinical study in which the participant is or will be exposed to an investigational or a non-investigational drug or device
* Medical status judged by study physician as contraindication

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos M Grilo, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale Department of Psychiatry, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yurkow S, Ivezaj V, Pittman B, Grilo CM. Preferences for Lisdexamfetamine vs Cognitive-Behavioral Therapy for Binge-Eating Disorder: Correlates and Outcomes. J Clin Psychiatry. 2025 May 7;86(2):24m15552. doi: 10.4088/JCP.24m15552. PMID 40338285

RESULTS

PARTICIPANT FLOW:
Groups:
- Lisdexamfetamine Dimesylate (LDX): Lisdexamfetamine Dimesylate: Participants randomly assigned to this arm will receive 12 weeks of LDX medication.
Period: Overall Study
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Cognitive-Behavioral Therapy | LDX and Cognitive Behavioral Therapy
Started | 47 | 47 | 47
Completed | 32 (Ten LDX participants stopped the treatment but completed the posttreatment assessment.) | 37 (One CBT participant completed treatment but not the posttreatment assessment.) | 35 (Ten LDX and Cognitive Behavioral Therapy participants stopped the treatment but completed the posttreatment assessment.)
Not Completed | 15 | 10 | 12
Not completed — Adverse Event | 10 | 0 | 10
Not completed — Withdrawal by Subject | 5 | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Cognitive-Behavioral Therapy | LDX and Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 47 | 47 | 47 | 141
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.85 (11.0) | 41.40 (12.59) | 44.0 (10.80) | 43.55 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 42 | 37 | 118
  Male | 8 | 5 | 10 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 7 | 4 | 19
  White | 36 | 36 | 35 | 107
  More than one race | 1 | 2 | 2 | 5
  Unknown or Not Reported | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 47 | 47 | 47 | 141

OUTCOME MEASURES:

1. Primary Outcome: Binge-Eating Frequency
Description: Binge eating will be assessed by interview and self-report and the primary outcomes is frequency. Frequency will be defined continuously (analyzed dimensionally).
Time Frame: Post-treatment (3 months)
Population: Any instance with a smaller N than specified in the participant flow table and footnote indicates a missing data point.
Measure: Mean (Standard Deviation); unit: Binge-eating episodes (past 28 days)
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Cognitive-Behavioral Therapy | LDX and Cognitive Behavioral Therapy
Number analyzed (Participants) | 42 | 36 | 45
Binge-eating episodes (past 28 days) | 2.95 (6.04) | 2.33 (5.88) | 0.96 (2.67)

2. Primary Outcome: Body Mass Index
Description: BMI is calculated using measured height and weight (e.g., percent loss). We note that % BMI change and % Weight Loss are exactly the same (when height is kept constant, which was the case with this short-term study with adults). Negative values indicate weight loss and positive values indicate weight gain.
Time Frame: Post-treatment (3 months)
Population: Any instance with a smaller N than specified in the participant flow table and footnote indicates a missing data point.
Measure: Mean (Standard Deviation); unit: percentage of change in weight
Groups:
- Lisdexamfetamine Dimesylate (LDX):: Lisdexamfetamine Dimesylate: Participants randomly assigned to this arm will receive 12 weeks of LDX medication.
Arm/Group | Lisdexamfetamine Dimesylate (LDX): | Cognitive-Behavioral Therapy | LDX and Cognitive Behavioral Therapy
Number analyzed (Participants) | 42 | 36 | 45
percentage of change in weight | -5.49 (3.47) | -0.50 (2.70) | -4.76 (3.57)

3. Secondary Outcome: Binge-Eating Remission
Description: Categorical: zero binges/28 days
Time Frame: Post-treatment (3 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Cognitive-Behavioral Therapy | LDX and Cognitive Behavioral Therapy
Number analyzed (Participants) | 47 | 47 | 47
Participants | 19 | 21 | 33

4. Secondary Outcome: Eating-Disorder Psychopathology
Description: Eating-disorder psychopathology is a continuous variable as assessed by the global score of the Eating Disorder Examination/Eating Disorder Examination-Questionnaire. Scores range from 0-6 (0=no eating-disorder psychopathology; 6=severe eating-disorder psychopathology).
Time Frame: Post-treatment (3 months)
Population: Any instance with a smaller N than specified in the participant flow table and footnote indicates a missing data point.
Measure: Mean (Standard Deviation); unit: scores on a scale ranging from 0-6
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Cognitive-Behavioral Therapy | LDX and Cognitive Behavioral Therapy
Number analyzed (Participants) | 39 | 35 | 44
scores on a scale ranging from 0-6 | 1.62 (0.94) | 1.89 (0.97) | 1.07 (0.68)

5. Secondary Outcome: Depressive Symptoms
Description: Depressive symptoms is a continuous variable of depressive symptomatology as assessed by the self-report measure, the Beck Depression Inventory - Second Edition. Scores range from 0-63 (0=no depressive symptoms, 63=greater depressive symptoms).
Time Frame: Post-treatment (3 months)
Population: Any instance with a smaller N than specified in the participant flow table and footnote indicates a missing data point.
Measure: Mean (Standard Deviation); unit: scores on a scale ranging from 0-63
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Cognitive-Behavioral Therapy | LDX and Cognitive Behavioral Therapy
Number analyzed (Participants) | 37 | 35 | 43
scores on a scale ranging from 0-63 | 8.24 (7.57) | 10.97 (10.26) | 7.02 (7.39)

ADVERSE EVENTS:
Time Frame: Reported adverse events were only monitored and collected for those receiving pharmacologic treatment for the first month of treatment.
Description: Mortality and serious adverse events were assessed for all intervention groups but adverse events (e.g., side effects expected for the study medication, LDX) were assessed only for the medication groups (LDX and LDX+CBT).
Arm/Group | Lisdexamfetamine Dimesylate (LDX) | Cognitive-Behavioral Therapy | LDX and Cognitive Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47 | 0/47
Serious Adverse Events (participants affected / at risk) | 1/47 | 0/47 | 0/47
Other Adverse Events (participants affected / at risk) | 46/47 | 0/0 | 46/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lisdexamfetamine Dimesylate (LDX) (N=47) | Cognitive-Behavioral Therapy (N=47) | LDX and Cognitive Behavioral Therapy (N=47)
Bruxism (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lisdexamfetamine Dimesylate (LDX) (N=47) | Cognitive-Behavioral Therapy (N=0) | LDX and Cognitive Behavioral Therapy (N=47)
Decreased appetite (Gastrointestinal disorders) | 42 | NA | 35
Dry Mouth (General disorders) | 28 | NA | 26
Increased Energy (General disorders) | 26 | NA | 25
Feeling Jittery (General disorders) | 18 | NA | 16
Insomnia (General disorders) | 14 | NA | 16
Increased Heart Rate (Nervous system disorders) | 10 | NA | 9
Diarrhea (Gastrointestinal disorders) | 6 | NA | 6
Constipation (Gastrointestinal disorders) | 5 | NA | 4
Anxiety (Psychiatric disorders) | 2 | NA | 10
Itchy Skin (General disorders) | 2 | NA | 6
Excessive Sweating (Nervous system disorders) | 1 | NA | 6
Tingling Sensation (Nervous system disorders) | 1 | NA | 4
Racing Thoughts (Psychiatric disorders) | 1 | NA | 5
Nightmare (General disorders) | 1 | NA | 3
Mouth/throat Pain (General disorders) | 1 | NA | 3
Changes to Thought Patterns (Psychiatric disorders) | 1 | NA | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT03924193/Prot_SAP_002.pdf
  • Informed Consent Form (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT03924193/ICF_001.pdf